CLINICAL TRIAL: NCT00010231
Title: Phase I Study Of Oral, 1,25 Dihydroxycholecalciferol (Calcitriol) + Dexamethasone In Hormone-refractory Prostate Cancer
Brief Title: Calcitriol Plus Dexamethasone in Treating Patients With Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCI-99044; CDR0000068457 (Registry Identifier: PDQ (Physician Data Query)); PCI-IRB-990606
Record Dates: First submitted 2001-02-02; First posted 2003-06-06 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Calcitriol; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: calcitriol
Drug: dexamethasone

SUMMARY:
RATIONALE: Combining calcitriol with dexamethasone may increase the effectiveness of therapy by making cancer cells more sensitive to dexamethasone.

PURPOSE: Phase I trial to study the effectiveness of calcitriol combined with dexamethasone in treating patients who have prostate cancer that has not responded to previous hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of calcitriol administered alone and in combination with dexamethasone in patients with hormone-refractory prostate cancer.
* Determine the pharmacokinetics of calcitriol with and without dexamethasone in these patients.

OUTLINE: This is a dose-escalation study of calcitriol.

In the first stage of the study, cohorts of 3-6 patients receive escalating doses of oral calcitriol on days 1-3. Dose escalation continues until the maximum tolerated dose (MTD) is determined.

In the second stage, patients receive escalating doses of oral calcitriol on days 1-3 and a fixed dose of oral dexamethasone on days 0-4. Treatment continues weekly in the absence of disease progression or unacceptable toxicity. Dose escalation continues until the MTD is determined.

Six additional patients may receive calcitriol and dexamethasone at one dose level below the MTD determined in the second stage, to confirm the MTD.

The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate with progressing regional or metastatic disease despite primary hormonal therapy (bilateral orchiectomy, estrogen, or luteinizing hormone-releasing hormone (LHRH) therapy with or without simultaneous antiandrogen)
* Documented new lesions or rising PSA (at least 50% increase on 3 measurements more than 2 weeks apart) after prior antiandrogen or progestational agent, or other hormonal agent cessation

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,500/mm^3
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL
* SGOT less than 4 times upper limit of normal

Renal:

* Creatinine no greater than 1.8 mg/dL

Other:

* No uncontrolled diabetes mellitus
* Fertile patients must use effective double barrier contraception for at least 1 week before, during, and at least 2 weeks after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Concurrent epoetin alfa for anemia allowed

Chemotherapy:

* Not specified

Endocrine therapy:

* See Disease Characteristics
* At least 28 days since prior antiandrogens or progestational agents
* Concurrent testicular androgen suppression with an LHRH analog (leuprolide or goserelin) allowed in non-orchidectomized patients

Radiotherapy:

* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No concurrent bisphosphonates

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 1999-06; Primary Completion 2002-08 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
MTD of calcitriol (oral) administered for 3 days (Monday, Tuesday, Wednesday -MTW) weekly in men with hormone-refractory prostate cancer | 1 year
MTD of calcitriol (oral, MTW weekly + dexamethasone (oral, Sunday, Monday, Tuesday, Wednesday - SMTW) in men with hormone refractory prostate cancer | 1 year

SECONDARY OUTCOMES:
whether dexamethasone permits the administration of calcitriol without the development of hypercalcemia in patients who developed hypercalcemia while receiving calcitriol alone | 1 year
pharmacokinetics of calcitriol when given as a single agent and following 3 days of dexamethasone | 1 year
effects of calcitriol +/- dexamethasone on serum PTH, urinary calcium and MAPK activity and VDR expression in serum, urine and PBMs , respectively, in this patient population | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gurkamal S. Chatta, MD, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States